CLINICAL TRIAL: NCT01037517
Title: Open Label Phase II Trial of an Augmented Mobilization Strategy With Plerixafor (Mozobil®) in a Population at Risk for Poor Stem Cell Mobilization
Brief Title: Trial of an Augmented Mobilization Strategy With Plerixafor (Mozobil®) in a Population at Risk for Poor Stem Cell Mobilization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Dr. David Szwajcer, Hematologist/Oncologist, CancerCare Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCM-002
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Myeloma; Lymphoma
Keywords: Myeloma; Multiple Myeloma or Lymphoma Patients undergoing; mobilization for the purpose of autologous stem cell collection
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Neoplasms, Plasma Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Successful Mobilizers (Active Comparator): Successful Mobilizers are defined as having a peripheral blood CD34 > 10X106/L.
  Interventions: Other: Observation: Nonintervention
- Poor Mobilizers (Experimental): Poor Mobilizer are defined as patients who on Day -1 have a peripheral blood [CD34] ≤ 10 X106/L
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor will be administered at 23:00 of Day -1 to experimental subjects at a dose of 240 mcg/kg subcutaneously, and possibly repeated the following day
  Other Names: Mozobil®
  Arms: Poor Mobilizers
Other: Observation: Nonintervention — Nonintervention group, no drug will be given, observation only
  Arms: Successful Mobilizers

SUMMARY:
Poor mobilization of hematopoietic progenitors needed to support autologous transplantation is a serious clinical problem. We are investigating the role of plerixafor administered in an at risk population to augment successful stem cell collection.

OBJECTIVES

To determine if plerixafor when administered on the day prior to planned autologous collection on first mobilization attempt in those with a peripheral blood CD34 ≤ 10X106/L will:

* increase the number of patients successfully collected in one day
* increase the number of patients successfully mobilized on first collection attempt
* is cost neutral within a Canadian setting

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years of age or older
2. Patients must be able to provide written consent
3. Participants must have a diagnosis of lymphoma or multiple myeloma and be undergoing autologous stem cell mobilization for the purposes of ASCT
4. Females of child bearing age will be asked to use an approved form of contraception

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding
2. Patients whose creatinine ≥ 250 μM
3. Serum AST, ALT or total bilirubin >5X upper limit of normal
4. Acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To increase the proportion of Poor Mobilizers who after receiving plerixafor are successfully collected in one day. The anticipated proportion increase is from 30%-60%. | within 1-2 days after commencing therapy

SECONDARY OUTCOMES:
To increase the proportion of Poor Mobilizers who after receiving plerixafor are successfully collected on first mobilization attempt rather than requiring a second mobilization. | After therapy
To describe the kinetics of platelet and neutrophil recovery post ASCT in those treated and not treated with plerixafor | After therapy
To examine the immune recovery at day 100 post ASCT in those treated and not treated with plerixafor | After therapy
To undertake a pharmacoeconomic evaluation to examine the impact of plerixafor on resource utilization in a population at risk for poor mobilization | After therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Official CancerCare Manitoba Website — http://www.cancercare.mb.ca